CLINICAL TRIAL: NCT04802837
Title: A Randomized, Double Blind, Active Controlled Study to Evaluate the Safety and Tolerability of Ridinilazole Compared With Vancomycin and to Assess the Pharmacokinetics of Ridinilazole in Adolescent Subjects (Aged 12 to <18 Years) With Clostridioides Difficile Infection
Brief Title: Safety, Tolerability and the Pharmacokinetics of Ridinilazole in Adolescent Subjects
Acronym: Ri-CoDIFy 3
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: SMT19969-C006 study was terminated in alignment with corporate decision to pursue further development of drug candidate with a partner.
Sponsor: Summit Therapeutics (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMT19969/C006; HHSO100201700014C (Other: Department of Health and Human Services)
Record Dates: First submitted 2021-03-09; First posted 2021-03-17 (Actual); Results first posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-07

CONDITIONS: Clostridioides Difficile Infection
Keywords: Clostridioides difficile infection (CDI); ridinilazole; Adolescents; vancomycin; C. Diff; Clostridium difficile; Diarrhea; Infection; Pediatric
MeSH Terms: conditions — Clostridium Infections; Diarrhea; Infections | interventions — ridinilazole; Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ridinilazole (Experimental): Ridinilazole dosed BID and a comparator placebo dosed QID, to maintain blind, for 40 doses over 10 days.
  Interventions: Drug: Ridinilazole
- Vancomycin (Active Comparator): Vancomycin dosed QID and a Ridinilazole placebo dosed BID, to maintain blind, for 40 doses over 10 days.
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Ridinilazole — Ridinilazole 200mg dosed BID for 10 days.
  Arms: Ridinilazole
Drug: Vancomycin — Vancomycin 125mg dosed QID for 10 days.
  Arms: Vancomycin

SUMMARY:
Study to evaluate the safety of ridinilazole in adolescent subjects and how ridinilazole is metabolized.

ELIGIBILITY:
Inclusion Criteria:

* Is aged 12 to <18 years.
* Has signs and symptoms of CDI including diarrhea such that in the Investigator's opinion CDI antimicrobial therapy is required, and the subject has tested positive for toxin A and/or B of C. difficile in the stool. Diarrhea is defined as ≥ 3 unformed bowel movements (UBMs) based on types 5, 6, 7 on the Bristol Stool Chart and diarrhea information is within 24 hours prior to randomization.

Exclusion Criteria:

* Has had more than the equivalent of 48 hours of dosing of antimicrobial treatment active against the current episode of CDI prior to randomization.
* Has received ridinilazole or an investigational vaccine against C. difficile any time in the past, anti-toxic antibodies including bezlotoxumab within the past 6 months, or any other investigational medicinal product for treatment of CDI or fecal microbiota replacement therapy within the past 3 months.
* Has a clinically relevant positive stool test for pathogens other than C. difficile, within 48 hours of randomization.
* Has life-threatening or fulminant CDI with evidence of hypotension, septic shock, peritoneal signs or absence of bowel sounds, toxic megacolon, or ileus.
* Has had major GI surgery (e.g. significant bowel resection or pancreatectomy but not including appendectomy or cholecystectomy) within past 3 months or has the presence of a colostomy or ileostomy or has the likely requirement of an ostomy during the study.
* Is receiving treatment that generally is associated with severe diarrhea, intractable vomiting, severe nausea, or inability to swallow that cannot be managed with antiemetics or antidiarrheals and that limits the ability to take oral medications. Cancer treatment that does not comprise ability to take study medication or cause severe diarrhea is allowed.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2021-09-17 (Actual); Study Completion 2022-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori Styles, MD, Study Director — Summit Therapeutics
Locations (18):
- United States (18):
  - University of California, Los Angeles (UCLA) David Geffen School of Medicine, Los Angeles, California
  - Children's Hospital Orange County, Orange, California
  - Continental Clinical Research, Miami, Florida
  - Dynamic Medical Research LLC, Miami, Florida
  - D&H National Research Centers, Miami, Florida
  - HMD Research, Orlando, Florida
  - Children's Center for Digestive Health, Atlanta, Georgia
  - Snake River Research, Idaho Falls, Idaho
  - Ann and Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Chicago - Comer Children's Hospital, Chicago, Illinois
  - Indiana University Health - Riley Hospital for Children, Indianapolis, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - DiGiovanna Institute for Medical Education and Research, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center - Rainbow Babies and Children's Hospital, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ridinilazole | Vancomycin
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ridinilazole | Vancomycin | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence and Severity of Treatment-emergant Adverse Events
Description: Safety was assessed using CTCAE v4.
Time Frame: Until study completion (Day 100)
Population: No analysis was done for study outcome measures due to the fact that enrollment in the clinical trial did not reach the target number of subjects needed prior to study termination and was insufficient to produce statistically reliable results.
Measure: Count of Participants; unit: Participants
Arm/Group | Ridinilazole | Vancomycin
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Until study completion (Day 100)
Description: No adverse event was reported throughout the duration of the study.
Arm/Group | Ridinilazole | Vancomycin
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2021-11-12): https://cdn.clinicaltrials.gov/large-docs/37/NCT04802837/Prot_000.pdf